CLINICAL TRIAL: NCT00005417
Title: Fifteen Year Follow-up of 5,500 Black and 5,500 Other Hypertensives
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4335; R03HL047677 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Kidney Failure, Chronic
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Kidney Failure, Chronic

SUMMARY:
To seek predictors of mortality, hospitalization, and dialysis using data from a hypertensive population which began treatment in 1974.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Patients dying before 1989 were identified using the VA's Beneficiary Identification Records Location Subsystem and the National Death Index (NDI). Using NDI information to locate them, death certificates were obtained on all dead patients. Arrangements were made to collect data on the VA hospitalizations occurring after antihypertensive treatment had begun, and application was made to match patients against the USRDS Dialysis and Transplant Registry. The basic clinical data were collected in 32 VA Hypertension Screening and Treatment Program (HSTP) clinics during the 40 month period beginning in 1974. Approximately 30,000 completed Screening and Evaluation Forms and 75,000 Treatment Visit Forms were completed during the 40 months of data collection. The collected information was entered into the HSTP Master File at the VA Computer Center in Austin, Texas. Predictors were sought for (1) all-cause mortality, (2) cause-specific mortality (obtained from death certificates and hospitalization and clinic records), (3) endstage renal disease (obtained from the USRDS Dialysis and Transplant Registry), (4) VA hospital usage combined with other data related to cost care.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-09; Study Completion 1993-09 (Actual)

REFERENCES:
- [Background] Perry HM Jr, Miller JP, Fornoff JR, Baty JD, Sambhi MP, Rutan G, Moskowitz DW, Carmody SE. Early predictors of 15-year end-stage renal disease in hypertensive patients. Hypertension. 1995 Apr;25(4 Pt 1):587-94. doi: 10.1161/01.hyp.25.4.587. PMID 7721402